CLINICAL TRIAL: NCT01061775
Title: Effects of Exenatide on Hypothalamic Obesity
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0903-028
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Hypothalamic Obesity
Keywords: Hypothalamic Obesity; Exenatide; Byetta; Craniopharyngioma
MeSH Terms: conditions — Sexual Infantilism; Craniopharyngioma | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exenatide (Experimental): 5mcg of exenatide will be given twice a day for 4 weeks and increased to 10 mcg twice a day for 20 weeks.
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — 5mcg twice a day for 4 weeks increased to 10 mcg twice a day for 20 weeks.
  Other Names: Byetta

SUMMARY:
The primary aim of this study is to evaluate the effect of Exenatide on weight status (change in body mass index) of children treated for craniopharyngioma that have developed hypothalamic obesity at Children's Hospitals and Clinics of Minnesota. We hypothesize that Exenatide given to hypothalamic obese children for 6 months will reduce their body mass index significantly from baseline.

DETAILED DESCRIPTION:
Hypothalamic obesity is when individuals suffer from acute weight gain after brain tumor treatment, involving secondary damage to the ventromedial nucleus of the hypothalamus, which may lead to obesity. The weight gain is uncontrolled and not receptive to diet and exercise interventions. The rate of long-term obesity in children diagnosed with craniopharyngioma can be as high as 50%. Exenatide, a drug indicated for diabetes, is an incretin mimicking agent that mimics the enhancement of glucose-dependent insulin secretion and several other antihyperglycemic actions of incretins has resulted in weight loss when given to diabetics. Exenatide shows potential to benefit patients suffering from hypothalamic obesity by slowing gastric emptying and therefore reducing food intake. Also increasing the glucagon-like peptide 1 (GLP-1) circulation, decreased due to obesity, at the already compromised GLP-1 receptor site of the hypothalamus could potentially help with regulation of appetite.

ELIGIBILITY:
Inclusion Criteria:

* >/=6 months post surgical or radiation or chemotherapy treatment for 1° craniopharyngiomas or other suprasellar tumors
* 10-21 years old
* Age-and sex-adjusted BMI >/=95%
* Parent sign consent and patient sign assent

Exclusion Criteria:

* < 6 months post surgical or radiation or chemotherapy treatment for 1° craniopharyngiomas or other suprasellar tumors
* Pregnant or breastfeeding, or those women who plan to get pregnant
* Renal impairment
* Gastroparesis
* Pancreatitis
* Diabetes
* <1 month post initiation of Metformin treatment
* Prescription or over-the-counter weight loss medications within 3 months of screening
* Are actively participating in, or have participated in a formal weight loss program within the last 3 months
* Have had bariatric surgery

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2010-01; Primary Completion 2013-07 (Actual); Study Completion 2019-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Jennifer Abuzzahab, MD, Principal Investigator — Children's Hospitals & Clinics of Minnesota
Locations (2):
- United States (2):
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospitals & Clincis of Minnesota, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data.

REFERENCES:
- See also: Hospital website — http://www.childrensmn.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide: Participants received 5mcg of exenatide twice a day for 4 weeks and increased to 10 mcg twice a day for 20 weeks.
Period: Overall Study
Arm/Group | Exenatide
Started | 19
Completed | 16
Not Completed | 3
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Exenatide
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 15 [10 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 19
Tumor Type [Number; unit: participants]
  Craniopharyngioma | 14
  Optic chiasm-hypothalamic glioma | 2
  Suprarasellar germinoma | 2
  Thalamic astrocytoma | 1
BMI [Mean (Full Range); unit: kg/m^2] | 35 [26.9 to 45.8]
Height [Mean (Standard Deviation); unit: cm] | 160.8 (14.3)
Weight [Mean (Standard Deviation); unit: kg] | 89 (28.2)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 111.6 (19.5)
Hip Circumference [Mean (Standard Deviation); unit: cm] | 113.5 (16)
Waist to Height Ratio [Mean (Standard Deviation); unit: cm] | 0.98 (0.08)
Child Eating Behaviour Questionnaire [Mean (Full Range); unit: units on a scale] — The Child Eating Behaviour Questionnaire (CEBQ) was designed as parent-report measure comprised of 35 items, each rated on a five-point likert scale that ranges from never to always. We utilized the CEBQ as a self-report measure during this study; it has not been validated for such use. For the purposes of this study, we looked at the Satiety Responsiveness Subscale Scores (5 questions; total scores could range from 5-25 with lower scores denoting a lower level of satiety).
  units on a scale | 11.47 [5.0 to 16.0]

OUTCOME MEASURES:

1. Primary Outcome: BMI Change
Description: BMI was collected at baseline and 24 weeks
Time Frame: 24 weeks
Population: The effects of exenatide on BMI were analyzed using a paired t-test comparing BMI at baseline with BMI after six months of treatment with each patient serving as his or her own control.
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Exenatide
Number analyzed (Participants) | 16
kg/m^2 | -0.77 [-1.97 to 0.43]
Statistical Analysis 1: Comparison: Exenatide; Test type: Superiority or Other; p = .05, t-test, 2 sided

2. Primary Outcome: Waist to Height Ratio (WHtR)
Description: Waist circumference was measured at the natural waist level (midway between the lowest rib margin and the iliac crest) at baseline and 24 weeks
Time Frame: 24 weeks
Population: All analyses were performed using SPSS (version 20.0.0, SPSS Inc, Chicago, IL).
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Exenatide
Number analyzed (Participants) | 16
percentage | -2.06 (0.08)
Statistical Analysis 1: Comparison: Exenatide; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

3. Secondary Outcome: Childhood Eating Behavior Questionnaire (CEBQ)
Description: The Child Eating Behaviour Questionnaire (CEBQ) was designed as parent-report measure comprised of 35 items, each rated on a five-point likert scale that ranges from never to always. We utilized the CEBQ as a self-report measure during this study; it has not been validated for such use. For the purposes of this study, we looked at the Satiety Responsiveness Subscale Scores (5 questions; total scores could range from 5-25 with lower scores denoting a lower level of satiety). The results reported show the change between baseline and week 24 scores.
Time Frame: 24 weeks
Population: Paired t-tests were performed to compare the satiety survey (continuous). Three subjects discontinued prior to completing the Week 24 CEBQ.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Exenatide
Number analyzed (Participants) | 16
units on a scale | 14 [12.2167 to 15.7833]
Statistical Analysis 1: Comparison: Exenatide; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

4. Secondary Outcome: Calorie Intake Based on 3-day Diet Records
Description: Dietary data were collected via 3-day diet records (Crawford et al. 1994) twice during the study, at baseline and week 24. Three-day diet records were collected on consecutive days including one weekend day. A registered dietitian (RD) instructed subjects on dietary data collection at baseline appointment. Depending on the age and capacity of the subject, the patient, parent or a collaboration of both recorded dietary intake. A RD entered dietary data into Nutritionist Pro software (First DataBank, SanBruno, CA) and the mean difference was analyzed.
Time Frame: 24 weeks
Population: The sample size was small due to missing data
Measure: Mean (95% Confidence Interval); unit: kcals
Groups:
- Exenatide: Exenatide: 5mcg twice a day for 4 weeks increased to 10 mcg twice a day for 20 weeks.
  Of 55 potential participants screened, 19 agreed to participate. Reasons for decline included reluctance to add another medication to their current regimens, travel distance, and aversion to an injectable medication. Sixteen patients completed the study. Of the three who failed to complete the study, one was lost to follow up, and two dropped out due to difficulty adhering to the twice daily injections, but none experienced significant side effects from therapy. Three of the 19 patients were on chronic metformin therapy.
Arm/Group | Exenatide
Number analyzed (Participants) | 10
kcals | 406.700 [-117.088 to 930.488]
Statistical Analysis 1: Comparison: Exenatide; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Exenatide
Serious Adverse Events (participants affected / at risk) | 2/19
Other Adverse Events (participants affected / at risk) | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide (N=19)
cholecystitis (Endocrine disorders) | 2 (2) — 2 developed cholecystitis requiring cholecystectomy. Both super-responders, with 1 losing 18 lbs in six months and the other remaining on medication for a full year losing nearly 40 lbs. Both developed symptoms well after last dose of study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide (N=19)
Nausea and stomachache (Gastrointestinal disorders) | 14 (20)
vomiting (Gastrointestinal disorders) | 10 (20)
Diarrhoea (Gastrointestinal disorders) | 3 (6)
Abdominal Pain (Gastrointestinal disorders) | 4 (8)
Blood in Stool (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Reflux Gastritis (Gastrointestinal disorders) | 1 (1)
Absomen Sore to Touch (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (2)
Fatigue (General disorders) | 2 (2)
Injection Site Pain (General disorders) | 1 (1)
Body Aches (General disorders) | 2 (2)
Seasonal Allergies (Immune system disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3)
Ear Infection (Immune system disorders) | 2 (4)
Pharyngitis (Immune system disorders) | 2 (2)
Sinusitis (Immune system disorders) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Blood in Urine Present (Investigations) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes